CLINICAL TRIAL: NCT01789437
Title: Diameters and Wall-to-lumen Ratio of Retinal Arterioles in Patients With Retinal Vein Occlusion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Andrea Russo, Dr., Università degli Studi di Brescia
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DIAMETER-001
Record Dates: First submitted 2013-02-07; First posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Hypertensive Patients With Retinal Vein Occlusion
Keywords: retinal vein occlusion; systemic hypertension; arteriolar diameter
MeSH Terms: conditions — Retinal Vein Occlusion; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexamethasone Intravitreal Implant (Active Comparator)
  Interventions: Device: Dexamethasone Intravitreal Implant (Ozuredex)

INTERVENTIONS:
Device: Dexamethasone Intravitreal Implant (Ozuredex)

SUMMARY:
to evaluate the wall-to-lumen ratio (WLR) of retinal arterioles in hypertensive patients with retinal vein occlusion (RVO) before and after dexamethasone intravitreal implant 0.7 mg (DEX) compared to a matched control group of normal eyes in non-hypertensive subjects.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide written informed consent and comply with study assessments for the full duration of the study;
* age > 20 years;
* decreased visual acuity as a result of clinically detectable ME associated with either CRVO or BRVO;
* the duration of macular edema was required to be between 4 and 24 weeks for both CRVO and BRVO;
* retinal thickness in the central subfield (as measured using optical coherence tomography) had to be > 350 µm in the study eye.

Exclusion Criteria:

* the exclusion criteria were as follows: diabetes; previous intravitreal anti-VEGF therapy or intravitreal steroid therapy; previous photodynamic therapy or focal laser; active retinal or optic disc neovascularization; active or history of choroidal neovascularization; presence of rubeosis iridis; any active infection; glaucoma, current ocular hypertension, or a history of steroid-induced intraocular pressure (IOP) increase in either eye; or concurrent eye disease in the study eye that could compromise visual acuity (e.g., choroidal neovascularization, diabetic retinopathy, epiretinal membrane).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
change of outer arteriolar diameter | the primary endpoint was at 6 months
change of inner arteriolar diameter | the primary endpoint was at 6 months

SECONDARY OUTCOMES:
Secondary outcome measures were as follows: adverse ocular events; mean change in visual acuity; and mean change in central macular thickness. | Outcomes were analyzed at 4 intermediate time points: 30, 60, 90, and 150 days.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Russo, Dr., Principal Investigator — University of Brescia, Italy
Locations (1):
- Spedali Civili di Brescia, Brescia, BS, Italy